CLINICAL TRIAL: NCT06974890
Title: Effects of Shuttle Balance Training on Balance , Gait and Postural Control in Children With Mild Cognitive Impairment
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: REC/RCR& AHS/24/0744
Record Dates: First submitted 2025-04-24; First posted 2025-05-16 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Mild Cognitive Impairment
Keywords: Down syndrome; Shuttle balance training; Mild cognitive impairment; Pediatric balance scale; Berg balance scale
MeSH Terms: conditions — Cognitive Dysfunction; Down Syndrome

STUDY DESIGN:
Intervention Model Description: The study will be randomized controlled trial. Total __ subjects will be assigned by non probability convenient sampling technique. They were randomly assigned to experimental and control groups.
  The Berg balance scale, limits of stability test, GOAL test, Timed up and go tools will be used.
  Tests will be used as outcome measure tools for balance, walk, coordination and Physical activity.
  All measures will be taken at baseline and at the end of treatment session. The collected data will be analyzed in Statistical Package for the Social Sciences (SPSS) 25.0 version. If data will be normally distributed then parametric if not normally distributed than non-parametric test will be apply.
Who Masked: Participant
Masking Description: Participants will get separate treatment protocols and possible efforts will be put to mask the both group about the treatment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Shuttle Balance Training (Experimental): Shuttle balance training is a dynamic exercise program designed to improve balance, gait, and posture, especially beneficial for children with mild cognitive impairment. It includes activities like shuttle runs, lateral steps, single-leg balances, crossovers, figure-8 drills, obstacle courses, and reaction drills-all aimed at enhancing coordination, stability, and agility. The program typically runs for 45-minute sessions, three times a week. Pre-assessments are used to measure baseline abilities, and progress is monitored throughout. This type of training helps improve motor control, body awareness, and functional movement, leading to better balance, more stable gait, and improved postural control in daily activities.
  Interventions: Other: Shuttle Balance Training
- Baseline Treatment (Active Comparator): "Baseline treatment" refers to the standard or initial treatment that is provided to a patient.
  Baseline treatment sets a foundation for managing the patient's condition effectively. It ensures that the patient receives appropriate care based on current medical knowledge and guidelines, with the goal of improving health outcomes and quality of life. Duration of session will be 45 min and 3 sessions per week.
  * Control Group Considerations: Clarifying how participants assigned to the control group will receive standard care or placebo intervention to maintain ethical standards and enable comparison with the intervention group.
  * Outcome Measures: Specifying the outcome measures and assessment tools used to evaluate the effects of the intervention on balance, gait, and postural control, both immediately after the intervention period and potentially during follow-up assessments.
  Interventions: Other: Baseline Treatment

INTERVENTIONS:
Other: Shuttle Balance Training — Shuttle balance training is a form of dynamic balance exercise that uses a shuttle system-often a platform or track with resistance bands or gliders-to help improve stability, coordination, and strength. In children, this type of training plays a significant role in enhancing gait, balance, and posture by engaging core and lower limb muscles in controlled, functional movements. It encourages proprioceptive development, helping children become more aware of their body's position in space, which is crucial for maintaining upright posture and walking efficiently. Through repetitive and playful activities, shuttle balance training can aid in correcting abnormal gait patterns, improving postural alignment, and boosting confidence in physical activities.
  Arms: Shuttle Balance Training
Other: Baseline Treatment — Baseline treatment sets a foundation for managing the patient's condition effectively. It ensures that the patient receives appropriate care based on current medical knowledge and guidelines, with the goal of improving health outcomes and quality of life. Duration of session will be 45 min and 3 sessions per week.
  Control Group Considerations: Clarifying how participants assigned to the control group will receive standard care or placebo intervention to maintain ethical standards and enable comparison with the intervention group.
  Arms: Baseline Treatment

SUMMARY:
This study aims to investigate the impact of Shuttle Balance Training (SBT) on balance, gait, and postural control among children diagnosed with mild cognitive impairment (MCI). Mild cognitive impairment in children often manifests as challenges in cognitive processing, motor coordination, and daily activities that involve balance and movement. The research will employ a randomized controlled trial (RCT) design, involving children aged 6-12 years diagnosed with MCI.

Participants will be randomly assigned to either an experimental group receiving Shuttle Balance Training or a control group receiving standard care or placebo interventions. The Shuttle Balance Training protocol consists of structured sessions focusing on dynamic balance exercises, coordination drills, and proprioceptive challenges using shuttle devices. Training sessions will be conducted thrice weekly over a period of 12 weeks, with each session lasting approximately 45 minutes. The study will be randomized controlled trial. Total __ subjects will be assigned by non probability convenient sampling technique. They were randomly assigned to experimental and control groups. The Berg balance scale, limits of stability test, GOAL test, Timed up and go tools will be used. Tests will be used as outcome measure tools for balance, walk, coordination and Physical activity. All measures will be taken at baseline and at the end of treatment session. The collected data will be analyzed in Statistical Package for the Social Sciences (SPSS) 25.0 version. If data will be normally distributed then parametric if not normally distributed than non-parametric test will be apply.

DETAILED DESCRIPTION:
This study aims to investigate the impact of Shuttle Balance Training (SBT) on balance, gait, and postural control among children diagnosed with mild cognitive impairment (MCI). Mild cognitive impairment in children often manifests as challenges in cognitive processing, motor coordination, and daily activities that involve balance and movement. The research will employ a randomized controlled trial (RCT) design, involving children aged 6-12 years diagnosed with MCI.

Participants will be randomly assigned to either an experimental group receiving Shuttle Balance Training or a control group receiving standard care or placebo interventions. The Shuttle Balance Training protocol consists of structured sessions focusing on dynamic balance exercises, coordination drills, and proprioceptive challenges using shuttle devices. Training sessions will be conducted thrice weekly over a period of 12 weeks, with each session lasting approximately 45 minutes. The study will be randomized controlled trial. Total __ subjects will be assigned by non probability convenient sampling technique. They were randomly assigned to experimental and control groups.

The Berg balance scale, limits of stability test, GOAL test, Timed up and go tools will be used.

Tests will be used as outcome measure tools for balance, walk, coordination and Physical activity.

All measures will be taken at baseline and at the end of treatment session. The collected data will be analyzed in Statistical Package for the Social Sciences (SPSS) 25.0 version. If data will be normally distributed then parametric if not normally distributed than non-parametric test will be apply.

ELIGIBILITY:
Inclusion Criteria:

Children with mild cognitive impairment (50-70%IQ)

* Age group from 6 to 12 years
* Both male and female
* Children must have the physical and cognitive ability to engage in the activities
* Children should be in generally good health, without severe medical conditions or orthopedic issues

Exclusion Criteria:

* Children with severe cognitive impairment
* Children who have severe neurological disorders
* Children with visual and auditory impairment
* Children with severe sensory processing disorders

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Estimated)
Dates: Start 2025-04-15 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-07-10 (Estimated)

PRIMARY OUTCOMES:
Berg Balance Scale | Baseline , 4th week, 8th week & 12th week
  A scale that is used to determine the balance in an individual. It has total 14 items, It takes about 20 minutes to complete each item, which has a five-point ordinal scale from 0 to 4, where 0 represents the lowest level of function and 4 the most. It excludes the evaluation of gait.
  TOTAL SCORE (Maximum = 56)
Limits of Stability Test | Baseline , 4th week, 8th week & 12th week
  Limits of Stability (LoS) is a key measure for assessing dynamic balance and voluntary motor control by tracking changes in the center of mass (COM). It helps identify postural instability and fall risk by evaluating how far a person can lean or sway without losing balance. LoS Represents the max distance a person can sway intentionally in direction without losing their balance. Normal range is anteroposterior 12.5 degrees, and medio-lateral 16 degrees.
Goal-Oriented Assessment of Life skills (GOAL) Test | Baseline , 4th week, 8th week & 12th week
  A test of functional motor skills required for day-to-day functioning is the Goal-Oriented Assessment of Lifeskills (GOAL). The GOAL program, which is intended for children aged 7 to 17, includes seven enjoyable and inspiring activities that are based on real-life tasks that kids do on a daily basis. The 54 Steps-small units of clearly visible, useful conduct within the seven Activities-are the foundation for the GOAL scores. Three components of successful functional performance-accuracy, independence, and speed-are used to score these. Each Step is graded as pass or fail using the Record Form. The Fine Motor and Gross Motor Standard Scores and the Progress Score are then calculated by adding the Step scores.
The Timed up and Go test. | Baseline , 4th week, 8th week & 12th week
  The timed Up and Go test (TUG) is a relatively simple test used to assess a person's mobility and requires both static and dynamic balance. The patient sits on a standard armchair back against it and resting arm position, regular footwear is used, the patient walks to a line that is 3meters away turns around the line, walks back to the chair and sits down. When the patient's buttocks touches the seat, the test ends there. A stopwatch is used to measure the time. Higher time score indicates high fall risks and less functional independence.

CONTACTS AND LOCATIONS:
Overall Officials: ZAHRA AHMAD, MS-PPT, Principal Investigator — Riphah International University
Locations (1):
- Rising Sun Institute, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jelsma D, Geuze RH, Mombarg R, Smits-Engelsman BC. The impact of Wii Fit intervention on dynamic balance control in children with probable Developmental Coordination Disorder and balance problems. Hum Mov Sci. 2014 Feb;33:404-18. doi: 10.1016/j.humov.2013.12.007. Epub 2014 Jan 18. PMID 24444657